CLINICAL TRIAL: NCT07187206
Title: Safety and Efficacy of FETO in CDH Phase III
Acronym: CDH FETO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0362
Record Dates: First submitted 2025-08-21; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypoplasia; Pulmonary Hypertension
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Fetuses with severe or moderate congenital diaphragmatic hernia will be offered fetal tracheal occlu (Experimental): FETO balloon placement/removal
  Interventions: Device: FETO, Fetal Endoluminal Tracheal Occlusion
- Fetuses with severe or moderate congenital diaphragmatic hernia will receive standard of care and op (No Intervention): no intervention standard of care

INTERVENTIONS:
Device: FETO, Fetal Endoluminal Tracheal Occlusion — Fetal Endoluminal Tracheal Occlusion with Balloon placement for fetuses with congenital diaphragmatic hernia
  Arms: Fetuses with severe or moderate congenital diaphragmatic hernia will be offered fetal tracheal occlu

SUMMARY:
Tracheal occlusion IDE approved by FDA for congenital diaphragmatic hernia fetuses and standard of care control group

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate that the FETO procedure increases the neonatal survival to discharge and reduces long-term morbidity rates in fetuses found to have intrathoracic herniation of the liver with LCDH and o/e LHR < 30% or RCDH and o/e LHR < 45 % with intrathoracic liver herniation when compared to those that receive standard of care management that have comparable defects for side and fetal lung volumes estimates and intrathoracic liver herniation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women 18 years and older, who are able to consent
* Singleton pregnancy
* Gestational age at enrollment is prior to 296 weeks
* Intrathoracic liver herniation
* Isolated Left CDH with o/e LHR < 30% at enrollment (180 to 295 weeks) or
* Isolated Right CDH with o/e LHR < 45% at enrollment (180 to 295 weeks)
* Normal fetal karyotype with confirmation by culture results, CMA with non-pathological variants, WES or WGS. Results by fluorescence in situ hybridization (FISH) will be acceptable if the patient is > 26 weeks
* Cervical length by transvaginal ultrasound > 20 mm within 24 hours prior to FETO procedure
* Patient meets psychosocial criteria
* Informed consent understood

Exclusion Criteria

* Patient < 18 years of age
* Multi-fetal pregnancy
* History of natural rubber latex allergy
* Preterm labor, cervix shortened (< 20 mm at enrollment or within 24 hours prior to FETO balloon insertion) or uterine anomaly strongly predisposing to preterm labor, or placenta previa.
* Psychosocial ineligibility, precluding consent:

  * Inability to reside within 30 minutes of Cincinnati Children's Hospital Medical Center and inability to comply with the travel for the follow-up requirements of the trial.
  * The patient does not have a support person (e.g. spouse, partner, mother) available to stay with the patient for the duration of the pregnancy at Cincinnati Children's Hospital Medical Center.
* Bilateral CDH, isolated LCDH with o/e LHR ≥ 30%, isolated RCDH with o/e LHR > 45%, as determined by ultrasound.
* No liver herniation into thoracic cavity
* Additional fetal anomaly and chromosomal abnormalities, associated anomalies recognized to alter survival prognosis (i.e., congenital heart disease) or presence of an underlying genetic syndrome (i.e., Fryns) by ultrasound, MRI, or echocardiogram at the fetal treatment center.
* Maternal contraindication to fetoscopic surgery or severe maternal medical condition in pregnancy
* History of incompetent cervix with or without cerclage
* Placental abnormalities (previa, abruption, accreta) known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal HIV, Hepatitis-B, Hepatitis-C positive because of the increased risk of transmission to the fetus during maternal-fetal surgery. If the patient's HIV status is unknown, the patient must be tested and found to have negative results before enrollment.
* Positive Hepatitis B surface antigen or presence of Hepatitis C in maternal blood uterine anomaly such as Mullerian duct abnormality, large or multiple fibroids that prohibit safe fetoscopic procedure
* There is no safe or technically feasible fetoscopic approach to balloon placement
* Participation in another intervention study that influences maternal and fetal morbidity and mortality, or participation in this trial in a previous pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological female
Enrollment: 75 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2032-12-01 (Estimated); Study Completion 2033-03-01 (Estimated)

PRIMARY OUTCOMES:
Change lung growth on prenatal imaging | prenatal period up to 40 weeks gestation
  Change in o/eLHR and other prenatal imaging tests

SECONDARY OUTCOMES:
Change survival in the severe congenital diaphragmatic hernia subgroup in intervention group | 6 months
  change rate of survival

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center (CCHMC), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No